CLINICAL TRIAL: NCT06132191
Title: Expanded Access Use of Cemiplimab in Patients With Solid Tumors
Status: Approved for marketing | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R2810-Cemiplimab
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC); Basal Cell Carcinoma (BCC); Cutaneous Squamous Cell Carcinoma (CSCC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Basal Cell | interventions — cemiplimab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Cemiplimab
  Other Names: REGN2810

SUMMARY:
Provide expanded access of cemiplimab in patients with solid tumors

DETAILED DESCRIPTION:
Compassionate Use requests are only being considered in response to Individual Patient Investigational New Drug (IND) applications. Availability will depend on location.

Sex: All
Age Groups: Child, Adult, Older Adult